CLINICAL TRIAL: NCT04614584
Title: Phase 1 Safety-interaction Study of Mirtazapine for the Treatment of Methamphetamine Use Disorder
Brief Title: Mirtazapine and Methamphetamine Drug-drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director of Substance Use Research, San Francisco Department of Public Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20-30109
Record Dates: First submitted 2020-09-14; First posted 2020-11-04 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Methamphetamine Use Disorder; Drug Interaction; Cardiovascular Abnormalities
Keywords: Methamphetamine; Mirtazapine; Methadone; Drug Interaction
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Mirtazapine; Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirtazapine (Experimental): Mirtazapine 30 mg PO daily x 4 days
  Interventions: Drug: Mirtazapine; Drug: Methamphetamine
- Placebo (Placebo Comparator): Placebo 30 mg PO Daily x 4 days
  Interventions: Drug: Methamphetamine

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine 30 mg PO daily x 4 days
  Arms: Mirtazapine
Drug: Methamphetamine — Methamphetamine 30 mg IV once

SUMMARY:
This is a drug-drug interaction (DDI) study of mirtazapine for methamphetamine (MA) use disorder (MUD) to ensure the safety of this medication in the presence of a relevant dose of MA for people actively-using MA.

Aim 1: To determine if mirtazapine alters the cardiovascular response to IV MA.

Aim 2: To determine if the pharmacokinetics of IV MA are altered by mirtazapine administration.

Aim 3: To evaluate the above aims in the setting of concomitant administration of methadone.

This study involves two simultaneous within-subject drug-drug interaction studies, each comprised of 12 participants. A total of 24 subjects will be enrolled who have methamphetamine use disorder who will be classified into 2 groups: (Group 1: no opioids; Group 2: opioid use disorder on methadone maintenance). Subjects will be randomized to the order of mirtazapine and placebo (i.e. one-half will receive mirtazapine first, then placebo; one-half will receive placebo first, then mirtazapine).

DETAILED DESCRIPTION:
This is a drug-drug interaction (DDI) study of mirtazapine for methamphetamine (MA) use disorder (MUD) to ensure the safety of this medication in the presence of a relevant dose of MA for people actively-using MA. MA is a widely used psychostimulant associated with substantial morbidity and mortality. MA is more prevalent than many other drugs, including opioids, with 37 million users of MA and amphetamine worldwide and 1.4 million past-year users in the U.S. alone in 2016. The number of MA poisoning deaths has steadily risen in recent years, from >3,700 in 2014 to 10,333 in 2017. Importantly, MA has been recognized as contributing substantially to the U.S. opioid crisis, with about half of MA poisoning deaths also caused by opioids. In the U.S., the annual economic cost of MA use is estimated to be $23.4 billion and use is strongly associated with HIV transmission.

There are no FDA-approved pharmacologic treatments for MUD, a major gap in addiction medicine, especially because behavioral interventions alone have limited efficacy and would likely benefit from adjunctive pharmacologic therapy. Investigators' prior clinical trials included a Phase IIa trial (N=60) and a replication Phase IIb trial (N=120) demonstrating that mirtazapine (an adrenergic, serotoninergic, and dopaminergic generic medication currently approved to treat depression) 30mg orally once daily reduced MA use among MA-dependent men who have sex with men (MSM) and transgender women. Investigators were directed to conduct a DDI study to ensure the safety of mirtazapine with MA. This research is particularly relevant given the overlap of MA use disorder and opioid use disorder (OUD), which could raise additional safety concerns.

The primary objectives of this study are as follows:

1. To determine if mirtazapine 30mg daily alters the cardiovascular response to IV MA. The interaction of active medication (compared with placebo) with relevant doses of MA (30 mg) on cardiovascular (heart rate, blood pressure, QTc interval) parameters and adverse events, including serotonergic signs, will be assessed to gather safety information in the Phase I human laboratory.
2. To determine if mirtazapine alters the pharmacokinetics of IV MA. Pharmacokinetic parameters for MA and its major metabolites will be assessed over 48 hours under steady state mirtazapine (30 mg) or placebo, and relevant IV MA challenge (30 mg).
3. To evaluate the above aims in the setting of concomitant steady-state administration of morphine or methadone.

Design This study involves two simultaneous within-subject drug-drug interaction studies, each comprised of 12 participants. A total of 24 subjects will be enrolled who have MA use disorder who will be classified into 2 groups: (Group 1: no opioids; Group 2: opioid use disorder on methadone maintenance). Subjects will be randomized to the order of mirtazapine and placebo (i.e. one-half will receive mirtazapine first, then placebo; one-half will receive placebo first, then mirtazapine).

Procedures Screening assessments will be completed across two-to-four visits over 2 weeks. All screening assessments should be completed within 14 days after labs are drawn.

All subjects will complete the following study visits: screening 1 and 2, enrollment/admission to inpatient stay, 14-day inpatient stay, 14-day post-discharge follow-up visit.

After consent is obtained, eligibility will be determined over the following screening visits, including medical history and physical examination (including weight and height), review of systems, vital signs, concomitant medications, EKG, breathalyzer, labwork, SCID. Additional assessments will include the CDS-12, PSQI, TLFB for substance use, delayed discounting, BIS-11, Stroop Test, CUDIT-r, COWS, ACSA, BDI-II.

On the day of enrollment, study staff will confirm eligibility and transport patient to hospital for admission. Participant will receive a test infusion of MA 30mg IV. If participant tolerates test infusion within defined parameters, participant will be formally enrolled and randomized. First dose of study drug will be administered the evening of admission. On the fifth hospital day, participant will undergo MA challenge (single-blind placebo and 30mg IV for subjective, cardiovascular, and PK assessments). PK draws will continue for 48 hours after infusion.

Participant will begin the opposite condition on day 8 and complete the MA infusion procedures on day 12. After completion of PK studies on day 14, participant will be discharged.

A post-discharge safety check will be completed 10 days after discharge (+/- 7 days).

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking;
2. age 18-55 years inclusive;
3. meet DSM-V criteria for MA use disorder, as diagnosed via SCID;
4. provide MA-positive urine during screening;
5. have a resting heart rate of 50-90
6. have a systolic blood pressure ≤ of 100-150 mm Hg, and diastolic blood pressure of 45-90 Hg within two days prior to admission;
7. have a baseline EKG that demonstrates normal sinus rhythm, QTc < 440 msec in men or QTc < 450 msec in women;
8. have acceptable safety lab data, ALT / AST<3x upper limit nL; est GFR >50;
9. if female (except females of non-childbearing potential-e.g., at least 1 year post-menopausal or surgically sterile), not pregnant confirmed by negative pregnancy test nor lactating and willing to use a medically approved method of birth control to prevent pregnancy during the trial and for 7 days after the last dose of study medication.

10) For those who also use opioids and are on methadone maintenance treatment (Group 2), urine positive for methadone and negative for buprenorphine on admission.

Exclusion Criteria:

1. Have current cocaine, cannabis, or alcohol use disorder by DSM-V SCID;
2. current or past history of seizure disorder;
3. current ongoing treatment with psychotropic medications (e.g. antidepressants, antipsychotics, antiepileptics, sedative/hypnotics, narcotic analgesics);
4. urine positive for MA and other unplanned drugs on the day of admission and breathalyzer results negative for alcohol;
5. any prior adverse reaction to MA; including chest pain or epileptic seizure;
6. major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar illness but excepting stable major depressive disorder, generalized anxiety disorder, etc.) as assessed by the SCID;
7. have a current neurological disorder (e.g., organic brain disease, dementia) or medical condition which would make study compliance difficult or compromise informed consent;
8. history of suicide attempt(s) in the past 90 days or current suicidal intent or plan by SCID;
9. evidence of untreated or unstable serious medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease including active tuberculosis infection;
10. seeking treatment for MA problems at the time of the study;
11. any serious medical or psychiatric AE after test infusion of MA 30mg IV (e.g. sustained SBP>200 or DBP>100; sustained pulse >(220-0.85xAge).
12. any other circumstances that, in the opinion of the investigators, would compromise participant safety and/or successful completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Safety Measures | 24 Days
  QT interval associated with combined use of methamphetamine and mirtazapine with and without concomitant methadone use
Metabolism of methamphetamine in presence of steady state mirtazapine | 14 Days
  Metabolism of methamphetamine in combination with mirtazapine Pharmacokinetics of methamphetamine in combination with mirtazapine with or without concomitant methadone use

SECONDARY OUTCOMES:
Impact of mirtazapine on subjective effects of methamphetamine reinforcement | 14 Days
  Subjective effects questionnaire
Impact of mirtazapine on mood produced by methamphetamine use | 14 days
  Addiction Research Inventory short form
Urge for stimulant use in the presence of mirtazapine | 14 days
  Methamphetamine-based Questionnaire for Stimulant Urges
Preference for methamphetamine in the presence of mirtazapine | 14 days
  Drug Purchase Task
Impact of mirtazapine on discounting in the presence of methamphetamine | 14 days
  Delayed Discounting assessment

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Coffin, MD, MIA, Principal Investigator — Director, Substance Use Division, San Francisco Department of Public Health
Locations (3):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - San Francisco Department of Public Health, San Francisco, California
  - Substance Use Research Unit, San Francisco, California

IPD SHARING:
Plan to Share IPD: No